CLINICAL TRIAL: NCT03462719
Title: A Randomized, Open-label, Phase 3 Study of the Combination of Ibrutinib Plus Venetoclax Versus Chlorambucil Plus Obinutuzumab for the First-line Treatment of Subjects With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL).
Brief Title: A Study of the Combination of Ibrutinib Plus Venetoclax Versus Chlorambucil Plus Obinutuzumab for the First-line Treatment of Participants With Chronic Lymphocytic Leukemia (CLL)/Small Lymphocytic Lymphoma (SLL)
Acronym: GLOW
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108428; 2017-004699-77 (EudraCT Number); 54179060CLL3011 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-03-06; First posted 2018-03-12 (Actual); Results first posted 2022-03-28 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib; venetoclax; Chlorambucil; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Arm A: Ibrutinib and Venetoclax (I+VEN) (Experimental): Participants will initially receive ibrutinib (420 mg [milligrams]/day) for 3 cycles. Venetoclax dose ramp up (from 20 to 400 mg over 5 weeks) will begin at Cycle 4 and the combination of ibrutinib and venetoclax will be given for 12 cycles (each cycle is equivalent to 28 days). Participants who subsequently develop progressive disease may enter to Subsequent Therapy Phase to receive single-agent ibrutinib until disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax; Drug: Ibrutinib (as Subsequent Therapy)
- Treatment Arm B: Chlorambucil and Obinutuzumab (G-Clb) (Active Comparator): Participants will receive chlorambucil and obinutuzumab (G-Clb) for 6 cycles. Participants will receive obinutuzumab, 1000 mg intravenously (IV) on Days 1, 8 and 15 of Cycle 1, and on Day 1 of Cycles 2 to 6 and chlorambucil 0.5 milligrams per kilogram (mg/kg) body weight, on Days 1 and 15 of Cycles 1 to 6. Participants who subsequently develop progressive disease may enter to Subsequent Therapy Phase to receive single-agent ibrutinib until disease progression or unacceptable toxicity.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab; Drug: Ibrutinib (as Subsequent Therapy)

INTERVENTIONS:
Drug: Ibrutinib — Participants will receive ibrutinib 420 mg orally once daily up to 15 cycles.
  Arms: Treatment Arm A: Ibrutinib and Venetoclax (I+VEN)
Drug: Venetoclax — Participants will receive venetoclax in combination with ibrutinib for a total of 12 cycles, beginning at Cycle 4. For the first 5 weeks of venetoclax treatment, the treatment dose will be ramped up from 20 to 400 mg.
  Arms: Treatment Arm A: Ibrutinib and Venetoclax (I+VEN)
Drug: Chlorambucil — Participants will receive chlorambucil at a dose of 0.5 mg/kg body weight on Days 1 and 15 of Cycles 1 to 6.
  Arms: Treatment Arm B: Chlorambucil and Obinutuzumab (G-Clb)
Drug: Obinutuzumab — Participant will receive obinutuzumab 1000 mg intravenously on Days 1, 8, and 15 of Cycle 1, and Day 1 of Cycles 2 to 6.
  Arms: Treatment Arm B: Chlorambucil and Obinutuzumab (G-Clb)
Drug: Ibrutinib (as Subsequent Therapy) — Participants will receive ibrutinib 420 mg orally once daily until disease progression or unacceptable toxicity during the subsequent therapy phase.

SUMMARY:
The purpose of this study is to assess progression-free survival (PFS) from treatment with ibrutinib plus venetoclax (I+VEN) compared with obinutuzumab plus chlorambucil (G-Clb) as assessed by an Independent Review Committee (IRC).

ELIGIBILITY:
Inclusion Criteria:

* Adult participants who are: (a) greater than or equal to (>=) 65 years old or, (b) 18 to 64 years old and have at least 1 of the following:

  1. Cumulative Illness Rating Scale (CIRS) score > 6
  2. Creatinine clearance (CrCl) estimated less than (<) 70 milliliter per minute (mL/min) using Cockcroft-Gault equation
* Diagnosis of chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL) that meets International Workshop on Chronic Lymphocytic Leukemia (iwCLL) criteria
* Measurable nodal disease (by computed tomography [CT]), defined as at least one lymph node > 1.5 centimeter (cm) in longest diameter
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) Grade less than or equal to (<=) 2
* Active CLL/SLL requiring treatment per the iwCLL criteria

Exclusion Criteria:

* Prior anti-leukemic therapy for CLL or SLL
* Presence of deletion of the short arm of chromosome 17 (del17p) or known TP53 mutation detected at a threshold of >10 percent (%) variable allele frequency (VAF)
* Major surgery within 4 weeks of first dose of study treatment
* Known bleeding disorders (example, von Willebrand's disease or hemophilia)
* Central nervous system (CNS) involvement or suspected Richter's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2029-04-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (87):
- United States (3):
  - Norton Cancer Institute, Louisville, Kentucky
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Novant Health, Charlotte, North Carolina
- Belgium (5):
  - Institut - Jules Bordet, Anderlecht
  - ZNA Stuivenberg, Antwerp
  - Universitair Ziekenhuis Gent, Ghent
  - Virga Jessa Ziekenhuis, Hasselt
  - UZ Leuven Gasthuisberg, Leuven
- Canada (6):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Juravinski Cancer Centre, Hamilton, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - CIUSSS de l Est de l Ile de Montreal Installation Hopital Maisonneuve Rosemont, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
- Czechia (5):
  - Fakultni nemocnice Brno, Interni hematologicka a onkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Hemato-onkologicke oddeleni, Pilsen
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense C
  - Roskilde Sygehus, Roskilde
- France (9):
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - Hopital Claude Huriez, Lille
  - CHU Montpellier, Montpellier
  - Hopital Haut Leveque Service Maladie Du Sang, Pessac
  - Centre Hospitalier Universitaire de Reims, Hôpital Robert Debré, Reims
  - Institut Universitaire du Cancer Toulouse Oncopole, Toulouse
  - CHU Bretonneau, Tours
  - CHU-Nancy, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif
- Israel (6):
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Western Galilee Medical Center, Nahariya
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Netherlands (11):
  - Flevoziekenhuis, Almere Stad
  - OLVG, Amsterdam
  - Academic Medical Center, Amsterdam
  - Reinier de Graaf Gasthuis, Delft
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharinaziekenhuis, Eindhoven
  - Spaarne Gasthuis, Hoofddorp
  - Zuyderland Medical Center, Sittard-Geleen
  - Antonius hospital, Sneek
  - MC Haaglanden, The Hague
  - Elisabeth zkh, Tilburg
- Poland (5):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im M Kopernika w Lodzi, Lodz
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - Wojewodzki Szpital Specjalistyczny im Janusza Korczaka, Słupsk
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Russia (6):
  - Moscow Multidisciplinary Scientific and Clinical Center named after S P Botkin, Moscow
  - S.P. Botkin Moscow City Clinical Hospital, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Ryazan Regional Clinical Hospital, Ryazan
  - St.-Petersburg Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - FSBIFederal Centre of Heart, Blood and Endocrinology named after V.A.Almazov MoH of the RF, Saint Petersburg
- Spain (11):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hospital Clinico Universitario Salamanca, Salamanca
  - Hosp. Virgen Del Rocio, Seville
- Sweden (2):
  - Sunderby Sjukhus Medicinkliniken, Luelå
  - Karolinska Universitetssjukhuset Solna, Centrum för Hematologi, Stockholm, Stockholm
- Turkey (Türkiye) (5):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Ankara Universitesi Tip Fakültesi Ibn-i Sina Hastanesi, Ankara
  - Ondokuz Mayis University, Atakum
  - V K V Amerikan Hastanesi, Istanbul
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
- United Kingdom (8):
  - Birmingham Heartlands Hospital, Birmingham
  - Addenbrookes Hospital, Cambridge
  - Queen Mary University of London, Charterhouse Square
  - New Victoria Hospital, Glasgow
  - St James's Hospital, Leeds
  - Derriford Hospital, Plymouth
  - Barking Havering and Redbridge University Hospitals NHS Trust, Romford
  - Royal Hallamshire Hospital, Sheffield

REFERENCES:
- [Derived] Kater AP, Owen C, Moreno C, Follows G, Munir T, Levin MD, Benjamini O, Janssens A, Osterborg A, Robak T, Simkovic M, Stevens D, Voloshin S, Vorobyev V, Ysebaert L, Qin R, Steele AJ, Schuier N, Baeten K, Caces DB, Niemann CU. Fixed-Duration Ibrutinib-Venetoclax in Patients with Chronic Lymphocytic Leukemia and Comorbidities. NEJM Evid. 2022 Jul;1(7):EVIDoa2200006. doi: 10.1056/EVIDoa2200006. Epub 2022 May 13. PMID 38319255
- [Derived] Niemann CU, Munir T, Moreno C, Owen C, Follows GA, Benjamini O, Janssens A, Levin MD, Robak T, Simkovic M, Voloshin S, Vorobyev V, Yagci M, Ysebaert L, Qi K, Qi Q, Sinet P, Parisi L, Srinivasan S, Schuier N, Baeten K, Howes A, Caces DB, Kater AP. Fixed-duration ibrutinib-venetoclax versus chlorambucil-obinutuzumab in previously untreated chronic lymphocytic leukaemia (GLOW): 4-year follow-up from a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2023 Dec;24(12):1423-1433. doi: 10.1016/S1470-2045(23)00452-7. Epub 2023 Nov 6. PMID 37944541
- [Derived] Moreno C, Solman IG, Tam CS, Grigg A, Scarfo L, Kipps TJ, Srinivasan S, Mali RS, Zhou C, Dean JP, Szafer-Glusman E, Choi M. Immune restoration with ibrutinib plus venetoclax in first-line chronic lymphocytic leukemia: the phase 2 CAPTIVATE study. Blood Adv. 2023 Sep 26;7(18):5294-5303. doi: 10.1182/bloodadvances.2023010236. PMID 37315225

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm A (Ibrutinib + Venetoclax): Participants received ibrutinib 420 milligrams (mg) orally once daily for 3 cycles (each cycle is of 28 days) followed by the combination of ibrutinib 420 mg and venetoclax 400 mg orally once daily for 12 cycles (including a 5-week venetoclax dose ramp up starting in cycle 4). Participants who subsequently developed independent review committee (IRC)-confirmed progressive disease (PD) and had active disease requiring treatment were eligible to participate in the Subsequent Therapy Phase and received single-agent ibrutinib until disease progression or unacceptable toxicity.
- Treatment Arm B (Chlorambucil + Obinutuzumab): Participants received chlorambucil 0.5 milligrams per kilogram (mg/kg) body weight orally once daily on Days 1 and 15 of Cycles 1 to 6 in combination with obinutuzumab 1000 mgs intravenously (IV) once daily on Days 1, 8, and 15 of Cycle 1 and Day 1 of Cycles 2 to 6 (each cycle is of 28 days). Participants who subsequently developed IRC-confirmed progressive disease (PD) and had active disease requiring treatment were eligible to participate in the Subsequent Therapy Phase and received single-agent ibrutinib until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Started | 106 | 105
Completed | 15 | 30
Not Completed | 91 | 75
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Ongoing | 87 | 72

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab) | Total
Number analyzed (Participants) | 106 | 105 | 211
Age, Continuous [Mean (Standard Deviation); unit: years] | 71 (8.02) | 72 (6.16) | 71.5 (7.01)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 42 | 89
  Male | 59 | 63 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 101 | 99 | 200
  Unknown or Not Reported | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 101 | 101 | 202
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  BELGIUM | 7 | 2 | 9
  CANADA | 7 | 10 | 17
  CZECH REPUBLIC | 9 | 13 | 22
  DENMARK | 7 | 5 | 12
  FRANCE | 4 | 3 | 7
  ISRAEL | 6 | 12 | 18
  NETHERLANDS | 1 | 6 | 7
  POLAND | 12 | 10 | 22
  RUSSIAN FEDERATION | 23 | 16 | 39
  SPAIN | 10 | 9 | 19
  SWEDEN | 2 | 0 | 2
  TURKEY | 8 | 13 | 21
  UNITED KINGDOM | 8 | 4 | 12
  UNITED STATES | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: time between date of randomization and date of disease progression, as assessed by IRC, or date of death due to any cause, whichever occurs first, regardless of use of subsequent anti-cancer therapy prior to PD or death using iWCLL2008 criteria : New enlarged lymph nodes >15 mm, new hepatomegaly or splenomegaly, or other organ infiltrates, bone lesion, ascites or pleural effusion due to CLL; >=50% increase in longest diameter (LDi) from nadir in existing lymph node (LDi >15 mm) or >=50% increase from nadir in sum of diameters of multiple nodes (and at least 1 node with LDi >15 mm); >=50% increase from nadir in enlargement of liver/spleen; >=50% increase from baseline in lymphocyte count (ALC; to >=5*10^9/L); or >=50% increase from nadir in ALC in >=2 serial assessments if ALC is >=30000*10^9/L and lymphocyte doubling time is rapid unless considered treatment-related lymphocytosis; new cytopenia attributable to CLL; transformation to more aggressive histology.
Time Frame: Up to 2 years 10 months
Population: The intent-to-treat (ITT) analysis set included all randomized participants who were analyzed according to assigned treatment group, regardless of the actual treatment received.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Months | NA [31.24 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events. | 20.96 [16.59 to 24.67]
Statistical Analysis 1: Comparison: Treatment Arm A (Ibrutinib + Venetoclax) vs Treatment Arm B (Chlorambucil + Obinutuzumab); Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.216, 95% CI 2-sided [0.131 to 0.357]

2. Secondary Outcome: Minimal Residual Disease (MRD) Negative Rate
Description: MRD-negative rate is defined as the percentage of participants who achieved MRD-negative status (that is, less than [<] 1 chronic lymphocytic leukemia (CLL) cell per 10,000 leukocytes or <0.01 percentage [%]) in the bone marrow as assessed by next-generation sequencing (NGS). Participants with missing MRD data were considered MRD positive.
Time Frame: Up to 2 years 10 months
Population: The ITT analysis set included all randomized participants who were analyzed according to assigned treatment group, regardless of the actual treatment received.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Percentage of participants | 55.7 [46.2 to 65.1] | 21.0 [13.2 to 28.7]

3. Secondary Outcome: Complete Response Rate (CRR)
Description: Complete response rate is defined as the percentage of participants who achieved complete response or complete response with an incomplete marrow recovery (CRi) on or prior to initiation of subsequent anti-leukemic therapy per the IRC assessment. International Workshop on Chronic Lymphocytic Leukemia (iWCLL) 2008 criteria: CR- No lymphadenopathy and hepatosplenomegaly, no constitutional symptoms, neutrophils >1.5*10^9/liter (L), platelets >100*10^9/L, Hgb >11 gram per deciliter (g/dL), absolute lymphocyte count <4000/microliter (mcL) and normocellular bone marrow with <30% lymphocytes and no B lymphoid nodules; CRi- CR with incomplete recovery of bone marrow.
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Percentage of Participants | 38.7 [29.4 to 48.0] | 11.4 [5.3 to 17.5]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR: percentage of participants who achieved best overall response of either CR, CRi, nodular PR (nPR) and partial response (PR). iWCLL 2008 criteria: CR- No lymphadenopathy and hepatosplenomegaly, no constitutional symptoms, neutrophils >1.5*10^9/liter (L), platelets >100*10^9/L, Hgb >11 g/dL and ALC <4000/mcL, normocellular bone marrow with <30% lymphocytes and no B lymphoid nodules; CRi- CR with incomplete recovery of bone marrow; nPR- participants meet criteria for CR, but bone marrow biopsy shows B-lymphoid nodules (reflecting residual disease); PR-2 of following when abnormal at baseline: >=50% decrease in ALC, >=50% decrease in sum of products of multiple nodes, >=50% decrease in enlargement of spleen or liver; and 1 of following: neutrophils >1.5*10^9/L, Platelets >100*10^9/L and Hgb>11 g/dL or >=50% improvement over baseline in any of these; 50% reduction in bone marrow infiltrates or B lymphoid nodules; no new enlarged nodes or new hepatosplenomegaly.
Time Frame: Up to 2 years 10 months
Population: The ITT analysis set included all randomized participants who were analyzed according to assigned treatment group, regardless of the actual treatment received. Participants with missing post-randomization data were considered non-responders.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Percentage of participants | 86.8 [80.3 to 93.2] | 84.8 [77.9 to 91.6]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from date of randomization to date of death from any cause.
Time Frame: Up to 4 years 10 months
Population: The ITT analysis set included all randomized participants who were analyzed according to assigned treatment group, regardless of the actual treatment received. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 17 | 36
Months | NA [NA to NA] — Here "NA" indicates that median and 95% CI was not estimable due to insufficient number of events. | NA [NA to NA] — Here "NA" indicates that median and 95% CI was not estimable due to insufficient number of events.

6. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the interval between the date of initial documentation of a response including partial response with lymphocytosis (PRL) and the date of first documented evidence of PD or death or date of censoring per the IRC assessment. iWCLL 2008 criteria for PD: New enlarged nodes >1.5 cm, new hepatomegaly or splenomegaly, or other organ infiltrates; >= 50% increase from nadir in existing lymph node or >=50% increase from nadir in sum of product of diameters of multiple nodes; >=50% increase from nadir in enlargement of liver or spleen; >=50% increase from baseline in lymphocyte count (and to >=5*10^9/L) unless considered treatment-related lymphocytosis; new cytopenia (Hemoglobin b or platelets) attributable to CLL; transformation to a more aggressive histology.
Time Frame: Up to 2 years 10 months
Population: Population analyzed included ITT amongst who were responders (PR or better).
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 92 | 89
Months | 28.85 [28.68 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events. | 21.13 [15.93 to 25.10]

7. Secondary Outcome: Time-to-Next Treatment
Description: Time-to-next treatment was measured from the date of randomization to the start date of any subsequent anti-leukemic therapy.
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Months | NA [NA to NA] — Here "NA" indicates that median and 95% CI was not estimable due to insufficient number of events. | NA [31.54 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events.

8. Secondary Outcome: Time to Worsening as Measured by Using EuroQol 5 Dimension 5 Level Questionnaire (EQ-5D-5L)
Description: Time to worsening= time interval (months) from randomization to first observation of deterioration. EQ-5D-5L consists of a 5-item descriptive system and the EuroQol visual analog scale (EQ-5D VAS). EQ-5D-VAS self-rating records respondent's own assessment of his/her overall health status at time of completion, on scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Worsening is defined as a decrease of >= 7 points (on a 0-100 scale).
  EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe participant's current health state. Responses for 5 dimensions are combined into a 5-digit number describing respondents health state that can be converted into a single index value or utility score (using the United Kingdom weights), ranging from -1 to 1, where lower scores indicate a worse health status. Worsening is defined as a decrease of >=0.08 points (on a 0-1 scale).
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Months
  EQ-5D-5L: Visual Analogue Score | 8.34 [5.65 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events. | 24.18 [11.27 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.
  EQ-5D-5L: Utility Score | 14.29 [8.15 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events. | 24.11 [8.34 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.

9. Secondary Outcome: Time to Worsening Measured by European Organization for Research and Treatment of Cancer-Quality of Life Questionnaire (EORTC QLQ)-C30)
Description: Time to worsening= time interval from randomization to first observation of deterioration. EORTC QLQ-C30 includes 30 separate items: 5 functional scales (physical, role, emotional, cognitive, and social Functioning), 1 global health status (GHS) and QoL scale, 3 symptom scales (fatigue, nausea/vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). Each item, except GHS, is answered on 4-point scale (1=not at all to 4=very much) and GHS is measured on 1-7 scale: 1=very poor and 7=excellent. Scores derived using validated scoring algorithms as per EORTC QLQ-C30 Manual and linearly transformed in a range from 0-100. For functional and global QoL scales, higher scores=better level of functioning/QoL. For symptom-oriented scales, higher score=more severe symptoms. Worsening in functional and global health scores=decrease of >=10 points (on 0-100 scale) and in symptom scores=increase of >=10 points (on 0-100 scale).
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Months
  Global Health Status | 14.95 [8.38 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events. | 24.18 [13.86 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.
  Cognitive Functioning | 11.07 [5.95 to 24.05] | 14.03 [7.16 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.
  Emotional Functioning | NA [17.31 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events. | 25.00 [16.62 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events
  Physical Functioning | NA [19.42 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events. | NA [14.03 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events.
  Role Functioning | 11.10 [6.28 to 14.95] | 8.48 [5.62 to 16.69]
  Social Functioning | 11.10 [8.34 to 16.69] | 17.87 [11.07 to 25.30]
  Fatigue (Symptom Scale) | 8.38 [5.62 to 14.95] | 17.87 [8.44 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.
  Nausea/Vomiting (Symptom Scale) | 11.07 [8.28 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events. | NA [20.44 to NA] — Here "NA" indicates that median and upper limit of 95% CI was not estimable due to insufficient number of events.
  Pain (Symptom Scale) | 8.31 [5.45 to 13.90] | 11.01 [5.65 to 17.87]

10. Secondary Outcome: Time to Worsening and Time to Improvement as Measured by Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Total Score
Description: Responses to the 13-item FACIT Fatigue Scale are reported on a 5-point categorical response scale ranging from 0 (not at all) to 4 (very much). The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worst score) to 52 (best score). Time to Worsening is defined as time interval (months) from randomization to first observation of deterioration. Worsening is defined as a decrease >= 3 points (on a 0-52 scale). Time to improvement is defined as the time interval (months) from randomization to the first observation of improvement. Improvement is defined as an increase >=3 points (on a 0-52 scale).
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Months
  Time to Worsening | 8.15 [3.98 to 10.94] | 14.03 [8.61 to NA] — Here "NA" indicates that upper limit of 95% CI was not estimable due to insufficient number of events.
  Time to Improvement | 5.59 [3.81 to 11.20] | 3.75 [2.20 to 5.75]

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) as a Measure of Safety and Tolerability
Description: An adverse event (AE) is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: Up to 4 years 10 months
Population: The safety analysis set is defined as all randomized participants who received at least one dose of any one of the four study drugs (ibrutinib, venetoclax, chlorambucil, or obinutuzumab).
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Participants | 105 | 99

12. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Findings
Description: Number of participants with abnormal clinical laboratory findings (hematology and serum chemistry) were reported.
Time Frame: Up to 4 years 10 months
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Participants
  Hematology: Absolute Neutrophils Counts (Decrease) | 81 | 95
  Hematology: Hemoglobin (Decrease) | 38 | 42
  Hematology: Platelets (Decrease) | 52 | 78
  Hematology: Any hemoglobin, platelet, or ANC decrease | 94 | 103
  Chemistry: Alanine Transaminase (ALT) (Increase) | 22 | 26
  Chemistry: Aspartate Aminotransferase (AST) (Increase) | 23 | 30
  Chemistry: Alkaline Phosphatase (Increase) | 19 | 21
  Chemistry: Bilirubin (Increase) | 36 | 25
  Chemistry: Creatinine (Increase) | 33 | 17
  Chemistry: Creatinine Clearance (Decrease) | 40 | 17
  Chemistry: Hypercalcemia | 13 | 3
  Chemistry: Hypoalbuminemia | 36 | 20
  Chemistry: Hypocalcemia | 27 | 30
  Chemistry: Phosphate (Decrease) | 16 | 6
  Chemistry: Potassium (Decrease) | 25 | 9
  Chemistry: Potassium (Increase) | 31 | 22
  Chemistry: Sodium (Decrease) | 25 | 26
  Chemistry: Sodium (Increase) | 12 | 8
  Chemistry: Uric Acid (Increase) | 37 | 19

13. Secondary Outcome: Percentage of Participants With Sustained Hemoglobin Improvement
Description: Sustained hemoglobin improvement is defined as the percentage of participants who achieved an increase in hemoglobin levels from baseline by >= 2 grams per deciliter (g/dL) and lasts for at least 56 days without blood transfusion or growth factors.
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Percentage of Participants | 44.3 | 50.5

14. Secondary Outcome: Percentage of Participants With Sustained Platelet Improvement
Description: Sustained platelet improvement is defined as the percentage of participants who achieved an increase in platelet levels from baseline by >= 50% and lasts for at least 56 days without blood transfusion or growth factors.
Time Frame: Up to 2 years 10 months
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
Number analyzed (Participants) | 106 | 105
Percentage of Participants | 24.5 | 29.5

15. Secondary Outcome: Plasma Concentration of Ibrutinib and Venetoclax
Description: Plasma concentrations of ibrutinib and venetoclax were determined by validated liquid chromatography-tandem mass spectrometry.
Time Frame: Ibrutinib: Pre-dose-Day 1 of Cycles 2, 3, 5 and 6 (each cycle is defined as 28 days), Venetoclax: Pre-dose-Day 1 of Cycles 5 and 6
Population: The pharmacokinetics (PK) analysis set is defined as all randomized participants in Treatment Arm A who received at least one dose of ibrutinib and/or venetoclax and had at least one valid blood sample drawn for PK analysis. Here 'N' (number of participants analyzed) signifies number of participants who were evaluable for this endpoint. Here, "n (number analyzed)" is defined as number of participants analyzed for specified category.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax)
Number analyzed (Participants) | 79
Nanograms per milliliter (ng/mL)
  Ibrutinib: Pre-dose Day 1 Cycle 2 (Ibrutinib Alone): number analyzed (Participants) | 63
  Ibrutinib: Pre-dose Day 1 Cycle 2 (Ibrutinib Alone) | 5.70 (5.58)
  Ibrutinib: Pre-dose Day 1 Cycle 3 (Ibrutinib Alone): number analyzed (Participants) | 59
  Ibrutinib: Pre-dose Day 1 Cycle 3 (Ibrutinib Alone) | 6.20 (7.78)
  Ibrutinib: Pre-dose Day 1 Cycle 5 (Ibrutinib and Venetoclax): number analyzed (Participants) | 65
  Ibrutinib: Pre-dose Day 1 Cycle 5 (Ibrutinib and Venetoclax) | 6.37 (6.71)
  Ibrutinib: Pre-dose Day 1 Cycle 6 (Ibrutinib and Venetoclax): number analyzed (Participants) | 60
  Ibrutinib: Pre-dose Day 1 Cycle 6 (Ibrutinib and Venetoclax) | 5.90 (6.74)
  Venetoclax: Pre-dose Day 1 Cycle 5 (Ibrutinib + Venetoclax) | 1139 (959)
  Venetoclax: Pre-dose Day 1 Cycle 6 (Ibrutinib + Venetoclax): number analyzed (Participants) | 65
  Venetoclax: Pre-dose Day 1 Cycle 6 (Ibrutinib + Venetoclax) | 1765 (1573)

ADVERSE EVENTS:
Time Frame: Up to 4 years 10 months
Description: The safety analysis set is defined as all randomized participants who received at least one dose of any one of the four study drugs (ibrutinib, venetoclax, chlorambucil, or obinutuzumab).
Arm/Group | Treatment Arm A (Ibrutinib + Venetoclax) | Treatment Arm B (Chlorambucil + Obinutuzumab)
All-Cause Mortality (participants affected / at risk) | 17/106 | 36/105
Serious Adverse Events (participants affected / at risk) | 49/106 | 30/105
Other Adverse Events (participants affected / at risk) | 98/106 | 98/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A (Ibrutinib + Venetoclax) (N=106) | Treatment Arm B (Chlorambucil + Obinutuzumab) (N=105)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Acute Myocardial Infarction (Cardiac disorders) | 2 | 1
Angina Unstable (Cardiac disorders) | 1 | 0
Atrial Fibrillation (Cardiac disorders) | 7 | 0
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 3 | 0
Cardiac Failure Congestive (Cardiac disorders) | 0 | 1
Myocardial Infarction (Cardiac disorders) | 1 | 0
Sinus Node Dysfunction (Cardiac disorders) | 2 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Mesenteric Artery Thrombosis (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 2
Sudden Death (General disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis Chronic (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Gallbladder Rupture (Hepatobiliary disorders) | 0 | 1
Cytokine Release Syndrome (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 0
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Clostridium Colitis (Infections and infestations) | 1 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 0
Erysipelas (Infections and infestations) | 1 | 0
Escherichia Urinary Tract Infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumococcal Sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 6 | 6
Pneumonia Cytomegaloviral (Infections and infestations) | 1 | 0
Respiratory Tract Infection (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 3
Multiple Injuries (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound Necrosis (Injury, poisoning and procedural complications) | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Aspartate Aminotransferase Increased (Investigations) | 0 | 1
Blood Phosphorus Increased (Investigations) | 0 | 1
Neutrophil Count Decreased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 1
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Adenocarcinoma Gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myeloproliferative Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Ischaemic Stroke (Nervous system disorders) | 2 | 0
Spinal Cord Compression (Nervous system disorders) | 1 | 0
Toxic Encephalopathy (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0
Mental Disorder (Psychiatric disorders) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 0
Chronic Kidney Disease (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis Bullous (Skin and subcutaneous tissue disorders) | 1 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0
Pyoderma Gangrenosum (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Hypertensive Urgency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Venous Thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm A (Ibrutinib + Venetoclax) (N=106) | Treatment Arm B (Chlorambucil + Obinutuzumab) (N=105)
Anaemia (Blood and lymphatic system disorders) | 17 | 18
Leukopenia (Blood and lymphatic system disorders) | 1 | 6
Neutropenia (Blood and lymphatic system disorders) | 36 | 56
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 28
Atrial Fibrillation (Cardiac disorders) | 12 | 2
Palpitations (Cardiac disorders) | 6 | 3
Vertigo (Ear and labyrinth disorders) | 8 | 0
Abdominal Pain (Gastrointestinal disorders) | 2 | 5
Constipation (Gastrointestinal disorders) | 11 | 7
Diarrhoea (Gastrointestinal disorders) | 53 | 13
Dyspepsia (Gastrointestinal disorders) | 10 | 3
Mouth Ulceration (Gastrointestinal disorders) | 8 | 0
Nausea (Gastrointestinal disorders) | 28 | 27
Vomiting (Gastrointestinal disorders) | 15 | 14
Asthenia (General disorders) | 9 | 7
Chills (General disorders) | 2 | 12
Fatigue (General disorders) | 16 | 10
Oedema Peripheral (General disorders) | 15 | 3
Pyrexia (General disorders) | 6 | 18
Bronchitis (Infections and infestations) | 7 | 7
Conjunctivitis (Infections and infestations) | 7 | 2
Nasopharyngitis (Infections and infestations) | 4 | 7
Pharyngitis (Infections and infestations) | 6 | 1
Pneumonia (Infections and infestations) | 5 | 6
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 14
Urinary Tract Infection (Infections and infestations) | 17 | 4
Contusion (Injury, poisoning and procedural complications) | 5 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 28
Alanine Aminotransferase Increased (Investigations) | 3 | 5
Aspartate Aminotransferase Increased (Investigations) | 3 | 6
Neutrophil Count Decreased (Investigations) | 10 | 9
Weight Decreased (Investigations) | 8 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 5
Hyperphosphataemia (Metabolism and nutrition disorders) | 9 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 6 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 10 | 7
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 9 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6 | 8
Dizziness Postural (Nervous system disorders) | 4 | 6
Headache (Nervous system disorders) | 7 | 5
Insomnia (Psychiatric disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 6
Onychoclasis (Skin and subcutaneous tissue disorders) | 7 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5
Rash (Skin and subcutaneous tissue disorders) | 17 | 7
Haematoma (Vascular disorders) | 8 | 2
Hypertension (Vascular disorders) | 13 | 5
Hypotension (Vascular disorders) | 3 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2019-12-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT03462719/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/19/NCT03462719/SAP_001.pdf